CLINICAL TRIAL: NCT04599829
Title: Assessment of the Safety and Performance of Ankle Ligament Supports in the Context of a Return to Sport After Sprain
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision : Difficulties of inclusion and revision of the clinical evaluation report of the medical device under evaluation.
Sponsor: Decathlon SE (Industry)
Collaborators: EFOR, France (Industry)
Responsible Party: Sponsor
Other Study IDs: ankleSTRONG100-500-900
Record Dates: First submitted 2020-09-06; First posted 2020-10-23 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2022-09

CONDITIONS: Ankle Sprain 1St Degree; Ankle Sprain 2Nd Degree; Ankle Sprain 3Rd Degree

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Orthosis Group 1: Use of AnkleSTRONG100 device
  Interventions: Device: AnkleSTRONG100/500/900
- Control Group 1: Control Group of the AnkleSTRONG100 Orthosis Group - No use of the device
- Orthosis Group 2: Use of AnkleSTRONG500 device
  Interventions: Device: AnkleSTRONG100/500/900
- Control Group 2: Control Group of the AnkleSTRONG500 Orthosis Group - No use of the device
- Orthosis Group 3: Use of AnkleSTRONG900 device
  Interventions: Device: AnkleSTRONG100/500/900
- Control Group 3: Control Group of the AnkleSTRONG900 Orthosis Group - No use of the device

INTERVENTIONS:
Device: AnkleSTRONG100/500/900 — At least 30 patients (15 patients in the orthosis group and 15 patients in the control group) per device type (3 device types: Ankle STRONG 100/500/900) totalling 90 patients will be included. Patients included in the orthosis group will use the device during sports sessions while patients included in the control group will not use an ankle support device.
  Groups: Orthosis Group 1; Orthosis Group 2; Orthosis Group 3

SUMMARY:
Decathlon has developed Ankle STRONG products which are medical devices that must be positioned around the ankle to limit ankle sprain occurrence.

The Ankle STRONG devices cover a range of 3 products (Ankle STRONG 100/500/900). The differences between the devices is based on the strength of compression and the ankle maintain.

The objective of this multicentre study is to collect data on the related clinical complications and clinical outcomes of market-approved Decathlon Ankle STRONG products to demonstrate safety and performance of these devices in a real-world setting.

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged ≥ 18 years old
* Subject has a recent mild OR moderate OR serious ankle sprain
* The current condition of his/her ankle allows the subject to resume usual physical activity
* Subject has been informed and is willing to sign an informed consent form
* Subject is willing to comply with protocol requirements and return to the study center for all clinical evaluations and required follow-up (12 weeks)
* Subject is affiliated to the French social security regime

Non-inclusion Criteria:

* Subject has conditions that may interfere with his/her ability to understand protocol requirements, participate in scheduled visits, or provide his/her informed consent
* Subject has worn a support (ankle brace or articulated orthosis) since his/her recent injury
* Subject has resumed regular physical activity since his/her recent injury
* Subject has any medical condition that could impact the study at investigator's discretion
* Subject has a known hypersensitivity or allergy to the components of the device (polyamide, elastane, polyester, cotton)
* Adult subject to legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject with ankle sprain whose current condition of his/her ankle allows the subject to resume usual physical activity
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Functional score | 12 weeks of follow-up
  Comparison of the functional result (Karlsson Ankle Function Score, 0-100 points) between the baseline and last follow-up visit in each group (orthosis vs control), for each device model

SECONDARY OUTCOMES:
Confidence level | At baseline and 12 weeks of follow-up
  Gap in the confidence level (patient rated outcome with 6 questions, ranging from 0 to 100) related to physical activity, between the baseline and last follow-up visit in each group (orthosis vs control), for each device model
Ankle instability | At 4 weeks, 8 weeks and 12 weeks of follow-up
  Comparison of ankle instability, assessed through a numerical rating scale (NRS, ranging from 0 to 10), between the groups (orthosis vs control), for each device model
Ankle pain | At 4 weeks, 8 weeks and 12 weeks of follow-up
  Comparison of ankle pain, assessed through NRS (ranging from 0 to 10), between the groups (orthosis vs control), for each device model
Safety (adverse events) | 12 weeks of follow-up
  Comparison of adverse events rates between the groups (orthosis vs control), for each device model

CONTACTS AND LOCATIONS:
Overall Officials: Valérie WIECZOREK, Principal Investigator — Centre Hospitalier Universitaire de Lille
Locations (1):
- Centre Hospitalier Universitaire de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No